CLINICAL TRIAL: NCT02621853
Title: Clinical Validation of High Throughput Raman Fiber Optic Probe to Determine Hepatic Fat Content
Brief Title: Clinical Validation of a Raman Spectroscope to Determine Hepatic Fat Content
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is also study sponsor. Dr. Alwayn is leaving NSHA and Canada for a new appointment in Europe.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 002
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2022-10

CONDITIONS: Steatosis
Keywords: Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI+RAMAN (Other): Patients will undergo an MRI for assessment of the fat content of the liver. Then during surgery, their livers will be illuminated (for a few seconds) by Raman spectroscope (the device in question) to see if MRI findings correlate well with Raman spectroscopy findings.
  Interventions: Device: Raman spectroscopy of the liver

INTERVENTIONS:
Device: Raman spectroscopy of the liver — Liver will be illuminated by the Raman spectroscope optic probe in order to assess fat content

SUMMARY:
Fatty liver disease including liver steatosis (fat deposition) is a major health problem worldwide. It is considered pathological when fat accumulation exceeds 5% of the liver weight. Transplantation represents the ultimate treatment for end stage liver disease. However, the discrepancy between the demand for donor organs and their availability presents one of the greatest hurdles of liver transplantation. Therefore, extended criteria organs have to be considered to overcome this shortcoming. Hepatic steatosis is one of the most important criteria defining extended-criteria donor liver. In liver transplantation, 'severe' fat deposition in donor liver is a major cause of graft failure while 'mild' deposition is considered transplantable and 'moderate' deposition represents the gray zone and remains difficult to assess. Surgeons usually perform a hepatic steatosis assessment during liver donor surgery. However, this method is very subjective and difficult especially when inexperienced surgeons or trainees are concerned. Furthermore, it has recently been documented that the assessment of steatosis is challenging even in the hands of experienced surgeons. Theoretically, a better way to assess steatosis before organ procurement would be a non-invasive imaging technique. However, some of these techniques appear to lack the sensitivity to accurately quantify hepatic fat content while others are complex, expensive and inconvenient to use in the setting of organ procurement. Therefore, liver biopsy remains the reference for grading hepatic steatosis. In daily practice the assessment and quantification of steatosis by a pathologist during organ procurement is more complex related to the lack of availability of dedicated hepatopathologists outside of office hours and in smaller community hospitals. A simple and short technique is therefore required to assess liver steatosis before retrieval. We have recently demonstrated that Raman spectroscopy could provide an accurate, rapid and real-time assessment of hepatic fat content and correlated highly with the gold standard (i.e. histopathological assessment of liver sections) in an animal model of liver steatosis. The purpose of this study is to validate the use of Raman spectroscopy for quantitative assessment of hepatic steatosis. In the hands of the surgeons this device can provide an immediate, robust tool to assess the suitability of donor livers at the site of retrieval prior to liver transplantation.

DETAILED DESCRIPTION:
Currently there are three main methods reported to assess liver steatosis before deceased donor liver retrieval: Noninvasive imaging techniques, evaluation of a liver biopsy sample by an experienced pathologist and assessment by transplant surgeon.

Imaging techniques that are currently in use include ultrasonography (USG) , computerized tomography (CT) and magnetic resonance imaging (MRI). Although it has an acceptable level of sensitivity, USG does not provide reproducible quantitative information. It can be used in most centers but it is operator dependent. Likewise, the diagnostic performance of non-enhanced CT scan for the accurate quantification of steatosis is unreliable. MRI is highly sensitive and specific in diagnosing hepatic steatosis and it has been reported that fat quantification using a 3.0-T MRI can provide sufficient sensitivity to detect and quantify steatosis in live liver donor candidates. However, this complex technology limits its use in routine organ procurement.

The microscopic evaluation of a liver biopsy sample by an expert pathologist is the gold standard for steatosis assessment. The presence and type of steatosis can be determined by microscopic evaluation. The grade of steatosis can be determined according to the international standards.

Despite being gold standard, biopsies are recorded for only 23% of transplanted livers in United States. Since a pathologist is not always available at the time of procurement, many centers rely mainly on the assessment of steatosis and organ quality by the procurement surgeon (i.e. transplant surgeon). During this assessment the donor liver is evaluated according to parenchymal texture criteria such as degree of yellowness (normal, mild, moderate, severe) and degree of firmness (soft, normal; mild, moderate, severe). However, studies which investigated how accurately a transplant surgeon could predict hepatic steatosis concluded that these assessments could be significantly misleading even in experienced hands.

Since all these three methods have their limitations, there is a need for a convenient and simple technique to better assess hepatic fat content prior to transplantation. Raman spectroscopy is an inelastic light scattering technique that is sensitive to molecular vibrations, the symmetry and frequencies of which are unique to the type of atoms and their spatial arrangement. Sensitivity to these properties is the basis of its ability to provide a spectral fingerprint of molecules in the illuminated region. It has been used to detect amino acids, nucleotide bases, fatty acids, saccharides, primary metabolites and other constituents that form the protein, carbohydrates, fats and DNA/RNA of biological tissues. It is an attractive technology for bioanalysis because no sample preparation is needed.

Raman spectroscopy is currently under investigation for use in clinical settings and it is carried out mainly for diagnostic purposes. It is currently approved for use in Canada for skin cancer diagnosis.

There are a variety of different Raman spectroscopy systems. We have recently designed a high throughput Raman spectroscopy system which is smaller than the others, portable and robust. It enables in situ scans of tissue to be undertaken with very little experience required of the operator. This system uses 'near infrared (NIR) excitation wavelength to improve the penetration depth of the laser while reducing the possibility of tissue damage. It gives information in the form of Raman spectra, analysis of which gives a Principal Component (PC) score.

This specially designed system could accurately quantify steatosis in mice and rat livers. The PC scores exhibited a significant correlation with histopathological examination results. Since steatosis in human liver tissue exhibit changes similar to the left liver lobe of mice and rats, we concluded that this technique could be applied to the field of transplantation. Clinical validation and subsequent adoption of this technique can provide transplant specialists with a valuable tool to obtain real time information on the severity of hepatic steatosis to assess the likelihood of a successful outcome and reduce inadvertent organ discard rates.

OBJECTIVE The aim of this study is to validate Raman spectroscopy (by means of our specially designed high throughput fiber optic Raman system) in a clinical setting in assessment of hepatic fat content. The in vivo Raman spectra (PC scores) will be compared to the findings of a pre-operative imaging method (MRI-fat quantification) and the current gold standard, liver biopsy (i.e. histopathological assessment of the liver specimen).

SPECIFIC RESEARCH QUESTIONS

1. Can Raman spectroscopy utilizing a portable fiber optic system rapidly assess the fat content of the liver in situ in clinical setting? 2. Do Raman spectra (principal component scores) correlate well with the findings of MRI-fat quantification and histopathological assessment of the liver biopsy specimen? STUDY DESIGN: This study is conceived as a single-centre, prospective validation study.

METHODS Partial liver resection is the surgical removal of a portion of the liver. Most partial liver resections are performed for the treatment of hepatic neoplasms. Patients who will undergo an open partial liver resection surgery in our institution will be reviewed with the circle of care team and approached for consent if deemed suitable for this study.

A Nova Scotia Health Authority Research Ethics Board-approved informed consent form will be utilized in the consent discussion (run by the clinical fellow or the research associate- both of whom are investigators participating in this project) and patients will be provided time to read the document in full before being asked for a decision on participation. Patients who give their consent for the study will be assigned to the study group. Assignment process will continue until 25 patients are included.

Study participants will undergo a pre-operative MRI for fat quantification. They will be asked to fast for at least 8 hours prior to MRI. Fat quantification technique (proton density fat fraction technique) will be performed using the IDEAL pulse sequence, which has been Health Canada approved for assessment of hepatic fat fraction, on a 3.0-T MR unit (GE 750; GE Healthcare). An attending fellowship trained abdominal radiologist who is experienced in MR image interpretation will measure the hepatic fat fraction (FF) on FF maps, which will be generated automatically. The automatically calculated hepatic FF will be displayed as a percentage on a full scale of 0-100.

During the liver resection procedure a region of the specimen that is to be removed but not the actual lesion will be illuminated by the Raman spectroscope fiber-optic probe. The Raman spectra provided and recorded in real-time (within a few seconds) will subsequently be analyzed (principal component analysis). This analysis will provide a PC score.

Following the application of Raman spectroscopy the operative procedure will continue as planned. Histochemical stains, H&E (hematoxylin-eosin) and trichrome, are routinely used for the interpretation of liver specimens in our anatomic pathology laboratory. As a special stain Oil Red O will need to be used to demonstrate the presence and extent of the fat (i.e. fat quantification) in liver tissue. Since it can only be performed on frozen sections a frozen section will be obtained from the removed liver specimen section to allow for Oil Red O staining- specific for diagnosing and quantifying fat droplets. An attending pathologist who is blinded to the MRI findings will evaluate these sections and determine the grade of steatosis as per the international standards:

M0: no macrovesicular steatosis M1: mild focal macrovesicular steatosis (<30% hepatocytes are involved) M2: moderate, zonal macrovesicular steatosis (>30 and <60% hepatocytes involved) M3: severe, panlobular macrovesicular steatosis (>60% hepatocytes involved) Correlation analysis will be performed between hepatic FF percentages, PC scores and steatosis grades for each study participant. Study participants will be followed after the surgery according to our standard post-liver resection follow-up protocol without any deviations from the standard of care.

STATISTICAL ANALYSIS For statistical analysis, quantitative data will be expressed as means and standard deviations and qualitative data will be expressed as numbers. Linear regression will be performed between macrovesicular steatosis grade and hepatic FF percentages and PC scores. Receiver operating characteristics (ROC) curves will be generated for the PC scores and hepatic FF percentages to identify their ability predict the grade of macrovesicular steatosis. All statistical analysis will be performed with commercially available statistical software (XLSTAT 2014).

Personal health information will not be used for the conduct of this project. Code numbers will be assigned for each participant. A database which will be accessible only to the investigators will be stored in a secured computer (requiring password entry) in transplant office (Queen Elizabeth II Health Sciences Centre, Victoria General Site, 4th floor, Dickson Building, Room 4074). This database will include the code numbers of the participants and the data elements such as hepatic FF percentage, PC score and steatosis grade.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥18 years of age), female/male patients who will undergo an open partial liver resection surgery in our institution will be included

Exclusion Criteria:

Patients who are scheduled for a metastasectomy or wedge resection where the margin of normal liver that is expected to be removed is less than 1 cm will be excluded.

In addition, patients who have the following will be excluded:

* Visual and/or mental impairment
* Coagulation disorder
* Cardiac pacemaker and/or defibrillator
* Deep brain stimulator
* Bullets or gunshot pellets
* Cerebral aneurysm clips
* Cochlear implant
* Magnetic dental implants
* Drug infusion devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Grade of steatosis determined according to the international standards by histopathological assessment of the liver biopsy specimen | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian Alwayn, MD, Principal Investigator — Dalhousie University

REFERENCES:
- [Background] Rogier J, Roullet S, Cornelis F, Biais M, Quinart A, Revel P, Bioulac-Sage P, Le Bail B. Noninvasive assessment of macrovesicular liver steatosis in cadaveric donors based on computed tomography liver-to-spleen attenuation ratio. Liver Transpl. 2015 May;21(5):690-5. doi: 10.1002/lt.24105. PMID 25761371
- [Background] Vetelainen R, van Vliet A, Gouma DJ, van Gulik TM. Steatosis as a risk factor in liver surgery. Ann Surg. 2007 Jan;245(1):20-30. doi: 10.1097/01.sla.0000225113.88433.cf. PMID 17197961
- [Background] Wertheim JA, Petrowsky H, Saab S, Kupiec-Weglinski JW, Busuttil RW. Major challenges limiting liver transplantation in the United States. Am J Transplant. 2011 Sep;11(9):1773-84. doi: 10.1111/j.1600-6143.2011.03587.x. Epub 2011 Jun 14. PMID 21672146
- [Background] Durand F, Renz JF, Alkofer B, Burra P, Clavien PA, Porte RJ, Freeman RB, Belghiti J. Report of the Paris consensus meeting on expanded criteria donors in liver transplantation. Liver Transpl. 2008 Dec;14(12):1694-707. doi: 10.1002/lt.21668. PMID 19025925
- [Background] Yersiz H, Lee C, Kaldas FM, Hong JC, Rana A, Schnickel GT, Wertheim JA, Zarrinpar A, Agopian VG, Gornbein J, Naini BV, Lassman CR, Busuttil RW, Petrowsky H. Assessment of hepatic steatosis by transplant surgeon and expert pathologist: a prospective, double-blind evaluation of 201 donor livers. Liver Transpl. 2013 Apr;19(4):437-49. doi: 10.1002/lt.23615. Epub 2013 Mar 17. PMID 23408461
- [Background] Sirlin CB. Noninvasive imaging biomarkers for steatosis assessment. Liver Transpl. 2009 Nov;15(11):1389-91. doi: 10.1002/lt.21875. No abstract available. PMID 19877212
- [Background] Park SH, Kim PN, Kim KW, Lee SW, Yoon SE, Park SW, Ha HK, Lee MG, Hwang S, Lee SG, Yu ES, Cho EY. Macrovesicular hepatic steatosis in living liver donors: use of CT for quantitative and qualitative assessment. Radiology. 2006 Apr;239(1):105-12. doi: 10.1148/radiol.2391050361. Epub 2006 Feb 16. PMID 16484355
- [Background] Castera L. Non-invasive diagnosis of steatosis and fibrosis. Diabetes Metab. 2008 Dec;34(6 Pt 2):674-9. doi: 10.1016/S1262-3636(08)74603-2. PMID 19195629
- [Background] Hewitt KC, Ghassemi Rad J, McGregor HC, Brouwers E, Sapp H, Short MA, Fashir SB, Zeng H, Alwayn IP. Accurate assessment of liver steatosis in animal models using a high throughput Raman fiber optic probe. Analyst. 2015 Oct 7;140(19):6602-9. doi: 10.1039/c5an01080b. Epub 2015 Aug 26. PMID 26309909
- [Background] Yu H, Shimakawa A, McKenzie CA, Brodsky E, Brittain JH, Reeder SB. Multiecho water-fat separation and simultaneous R2* estimation with multifrequency fat spectrum modeling. Magn Reson Med. 2008 Nov;60(5):1122-34. doi: 10.1002/mrm.21737. PMID 18956464
- [Background] Bohte AE, van Werven JR, Bipat S, Stoker J. The diagnostic accuracy of US, CT, MRI and 1H-MRS for the evaluation of hepatic steatosis compared with liver biopsy: a meta-analysis. Eur Radiol. 2011 Jan;21(1):87-97. doi: 10.1007/s00330-010-1905-5. Epub 2010 Jul 31. PMID 20680289
- [Background] Bravo AA, Sheth SG, Chopra S. Liver biopsy. N Engl J Med. 2001 Feb 15;344(7):495-500. doi: 10.1056/NEJM200102153440706. No abstract available. PMID 11172192
- [Background] Deroose JP, Kazemier G, Zondervan P, Ijzermans JN, Metselaar HJ, Alwayn IP. Hepatic steatosis is not always a contraindication for cadaveric liver transplantation. HPB (Oxford). 2011 Jun;13(6):417-25. doi: 10.1111/j.1477-2574.2011.00310.x. Epub 2011 Apr 7. PMID 21609375
- [Background] Spitzer AL, Lao OB, Dick AA, Bakthavatsalam R, Halldorson JB, Yeh MM, Upton MP, Reyes JD, Perkins JD. The biopsied donor liver: incorporating macrosteatosis into high-risk donor assessment. Liver Transpl. 2010 Jul;16(7):874-84. doi: 10.1002/lt.22085. PMID 20583086
- [Background] Ji R, Li YQ. Diagnosing Helicobacter pylori infection in vivo by novel endoscopic techniques. World J Gastroenterol. 2014 Jul 28;20(28):9314-20. doi: 10.3748/wjg.v20.i28.9314. PMID 25071325
- [Background] von Rundstedt FC, Lerner SP. New imaging techniques for nonmuscle invasive bladder cancer. Curr Opin Urol. 2014 Sep;24(5):532-9. doi: 10.1097/MOU.0000000000000093. PMID 25051025
- [Background] Gao L, Wang Z, Li F, Hammoudi AA, Thrall MJ, Cagle PT, Wong ST. Differential diagnosis of lung carcinoma with coherent anti-Stokes Raman scattering imaging. Arch Pathol Lab Med. 2012 Dec;136(12):1502-10. doi: 10.5858/arpa.2012-0238-SA. PMID 23194042
- [Background] Almond LM, Barr H. Advanced endoscopic imaging in Barrett's oesophagus. Int J Surg. 2012;10(5):236-41. doi: 10.1016/j.ijsu.2012.04.003. Epub 2012 Apr 14. PMID 22510441
- [Background] Hughes OR, Stone N, Kraft M, Arens C, Birchall MA. Optical and molecular techniques to identify tumor margins within the larynx. Head Neck. 2010 Nov;32(11):1544-53. doi: 10.1002/hed.21321. PMID 20091681
- [Background] Schaar JA, Mastik F, Regar E, den Uil CA, Gijsen FJ, Wentzel JJ, Serruys PW, van der Stehen AF. Current diagnostic modalities for vulnerable plaque detection. Curr Pharm Des. 2007;13(10):995-1001. doi: 10.2174/138161207780487511. PMID 17430163
- [Background] DaCosta RS, Wilson BC, Marcon NE. Optical techniques for the endoscopic detection of dysplastic colonic lesions. Curr Opin Gastroenterol. 2005 Jan;21(1):70-9. PMID 15687888
- [Background] Lui H, Zhao J, McLean D, Zeng H. Real-time Raman spectroscopy for in vivo skin cancer diagnosis. Cancer Res. 2012 May 15;72(10):2491-500. doi: 10.1158/0008-5472.CAN-11-4061. Epub 2012 Mar 20. PMID 22434431
- [Background] Markin RS, Wisecarver JL, Radio SJ, Stratta RJ, Langnas AN, Hirst K, Shaw BW Jr. Frozen section evaluation of donor livers before transplantation. Transplantation. 1993 Dec;56(6):1403-9. doi: 10.1097/00007890-199312000-00025. PMID 7506453